CLINICAL TRIAL: NCT02861677
Title: Impact of Clinical Pharmacy Service on Patient Care and Cost Saving
Acronym: TGPIONEER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jimma University (Other)
Collaborators: MSH/SIAPS-Ethiopia (Unknown)
Responsible Party: Principal Investigator, Tigestu Alemu, Lecturer and clinical pharmacist, Jimma University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Rpge/502/2016
Record Dates: First submitted 2016-08-01; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Health Care Improvement
MeSH Terms: interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group will receive the usual medical care by physicians and nurses
- Intervention group (Experimental): the intervention group will receive clinical pharmacy services
  Interventions: Other: pharmaceutical care

INTERVENTIONS:
Other: pharmaceutical care
  Arms: Intervention group

SUMMARY:
Background: Pharmacists have been proven to improve patient outcomes, medication adherence, glycemic control, reduce blood pressure, low-density lipoprotein, health care costs and length of hospital stay, and enhance quality of life.

Objective: to measure the impact of clinical pharmacy service on patient care and cost saving of patients at inpatient wards and ambulatory care clinics of Jimma University Specialized Hospital.

Methods: single center Randomized Controlled Trial will be conducted. Participants will be assigned to either pharmacy professionals' intervention group or non-intervention (control) group based on computer generated random number. The study will be done from July 26 to September 15, 2016. The total sample size is calculated with Open Epi online sample size calculator with 95% CI and 80% power. The total sample size is found to be 146 for inpatients and 473 for outpatients. Linear regression, student's t-test, logistic regression and chi-square test will be used for statistical analysis. Variables with p<0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
Many studies have shown the positive impact of clinical pharmacy service on clinical, economic and humanistic outcomes. This type of service may be highly important in saving lives, improving patient outcomes, and decreasing treatment costs particularly in resource-limited settings like Ethiopia with a double burden of communicable and non-communicable diseases which need medication therapy. Though patients may experience a number of problems related to drug therapy, no study is conducted in Ethiopia to show the impact of clinical pharmacy service in alleviating such treatment related problems.

Therefore, this study aims to answer the following research questions.

impact of clinical pharmacy service in improving patient outcome and reducing cost of treatment of chronic illness patients

impact of clinical pharmacy service in improving patient outcome and reducing cost of treatment of hospitalized patients

Study site location and participants: this randomized controlled trial will be conducted at Jimma University Specialized Hospital, Southwest Ethiopia.

Sample size calculation

The sample size for inpatients is calculated using the Open Epi online sample size calculator software with the following assumptions:

With 80% power and significance level of 0.05 with a 95% confidence interval. Two tailed test and a 1:1 ratio between intervention group and control group. The investigators used the prevalence of drug related problem (primary outcome) to be 52% from previous reports in Ethiopia.

The effect size is considered to be 1.5

Through calculation, the final sample size in each arm is 61 and considering a 20% contingency for loss to follow up, 73 participants are needed in each group. Therefore, the total sample size is 146.

For ambulatory patients, sample size is calculated using the prevalence of the three types of drug related problems (indication, safety, and effectiveness) from previous studies. The prevalence of effectiveness related drug related problem was reported to be 14%. The effect size is determined to be 1.4 and all other parameters are considered similar to the above. Through calculation, 215 patients are needed in each group. Considering a 10% loss for follow up, the total sample size is 473 in the two groups.

Randomization and concealing allocation

Randomization will be completed by Statistical Package for the Social Science version 21 generated algorithm. Treating assignments kept in sealed opaque envelopes with only number labeled will be opened after patients give their informed consents. The assigned research assistant will distribute envelopes and record patients in each group enrollment and patient assignment.

Blinding: research assistants of the trial who are responsible for outcome recording will be blinded to treatment assignment.

Intervention:

Pharmacy Intervention group

For Hospitalized Patients:

Four full timer pharmacists trained on clinical pharmacy (ward Pharmacists) will be assigned to 8-15 patients each at medical ward to provide clinical pharmacy service.

Two full timer postgraduate year two clinical pharmacy students will be assigned to medical ward A Male and medical ward B female.

Two clinical pharmacists from school of pharmacy will also be assigned to each ward.

For Ambulatory Patients;

Two post graduate year II clinical pharmacy students will be assigned to outpatient department of ambulatory care clinic.

The assigned pharmacy professionals will sit with the physician and make therapeutic decisions in consultation with the physician, develop therapeutic plan and give patient education and document into the documentation form.

Control Group

Patients in the control group will get the standard care by physicians and nurses.

Measurement

Primary outcomes

Interventions by Pharmacy professionals

For hospitalized patients, all interventions made by pharmacy professionals will be documented on pharmacy professional activity documentation forms. Data collectors will abstract all the relevant data from the document. The data that will be abstracted by data collectors are:

Identified drug therapy problems and interventions made to resolve drug therapy problems.

Suggestions on prevention and avoidance of medication errors.

Cost of medicines and pharmaceuticals.

Cost of hospitalization including cost of laboratory investigations.

Patient educations given during hospital stay and at discharge for hospitalized patients.

Recommendations made for laboratory investigation and treatment monitoring done.

Patient education at hospital for ambulatory patients.

Secondary outcomes

Length of hospital stay

In hospital mortality

Patient knowledge about the drug at discharge

Inpatient satisfaction with the health care service provided

For ambulatory patients,

Primary outcome

Identified drug therapy problems and interventions made to resolve drug therapy problems.

Cost of medicines

Secondary outcomes

Patient knowledge about the prescribed medicines

Statistical analysis: Statistical software Statistical Package for the Social Science 21 will be used for analysis. Variables with p value<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old,
* Patients admitted to internal medicine ward,
* Ambulatory patients with the following non-communicable diseases:

  * diabetes mellitus,
  * hypertension,
  * heart failure,
  * ischemic heart disease,
  * rheumatoid heart diseases,
  * chronic kidney disease,
  * venous thromboembolism,
  * asthma, chronic obstructive pulmonary disease, and epilepsy who have been on treatment for at least three months.

Exclusion Criteria:

* Hospitalized medical inpatients with the following conditions.
* Drop outs:

  * Patients leaving against medical advice, die and abscond within 72 hours of admission.
  * Patients not willing to participate.
  * Patients who may be transferred from intensive care unit to internal medicine ward.
  * Patients who may be transferred from other wards to internal medicine ward.
  * Patients admitted with stroke.

Chronic illness ambulatory patients with the following conditions:

* Patients not willing to participate.
* Women with gestational diabetes.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The number of drug therapy problems | through study completion, an average of 8 weeks
The number of medication errors | through study completion, an average of 8 weeks
Cost of medicines | through study completion, an average of 8 weeks

SECONDARY OUTCOMES:
Length of hospital stay | through study completion, an average of 8 weeks
In hospital mortality | through study completion, an average of 8 weeks

IPD SHARING:
Plan to Share IPD: No